CLINICAL TRIAL: NCT06037083
Title: Post-Extubation Assessment of Clinical Stability in Extremely Preterm Infants: the PEACE Feasibility Study
Brief Title: Post-Extubation Assessment of Clinical Stability in ELBW Infants
Acronym: PEACE
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Wissam Shalish, Assistant Professor of Pediatrics, McGill University Neonatologist, Montreal Children's Hospital, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-8794
Record Dates: First submitted 2023-09-01; First posted 2023-09-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Extremely Low Birth Weight Infants
Keywords: Reintubation; Extubation; Extremely low birth weight infants; Electrical impedance tomography; Cerebral and splanchnic oxygenation; Near infrared spectroscopy; apnea; intermittent hypoxia
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- 20 extremely low birth weight infants: In addition to the standard care, all participants will be monitored using an extra oxygen saturation probe, two near infrared spectroscopy sensors, and an electrical impedance tomography belt. Data will be continuously collected from extubation to 168 hours postextubation
  Interventions: Device: Oxygen saturation probe; Device: Near infrared spectroscopy sensors; Device: Electrical impedance tomography

INTERVENTIONS:
Device: Oxygen saturation probe — The high-accuracy oxygen saturation signal will be continuously acquired for 168 hours post extubation from a separate pulse oximeter (Radical-7®, Masimo ROOT platform, MasimoCorp, Irvine, LA).
Device: Near infrared spectroscopy sensors — The cerebral and splanchnic regional oxygen saturation signals will be acquired continuously for 168h post extubation using two near infrared spectroscopy sensors (Masimo ROOT platform, MasimoCorp, Irvine, LA), one placed on the forehead for cerebral oxygenation and one on the abdomen (for splanchnic oxygenation).
Device: Electrical impedance tomography — The regional lung ventilation will be measured using Electrical Impedance Tomography (TIMPEL, USA) at three time points:
  * From 1 hour pre-extubation to 2 hours post extubation (total 3 hours)
  * Between 24 and 48 hours post extubation (total 3 hours)
  * Between 72 and 96 hours post extubation (total 3 hours)

SUMMARY:
This is an observational, proof-of-concept, feasibility study that aims to evaluate the feasibility of a monitoring system that integrates clinical data, high-resolution waveforms from the bedside monitor, regional oxygenation (via cerebral and splanchnic near-infrared spectroscopy), and regional ventilation (via electrical impedance tomography) from 20 extremely low birth weight infants at high-risk of reintubation.

DETAILED DESCRIPTION:
The primary aim of this proof-of-concept study is to evaluate the feasibility and acceptance of a monitoring system that integrates clinical data and biomedical signals from multiple modalities in a cohort of extremely preterm infants at high-risk of clinical instability on non-invasive respiratory support.

Secondary aims will be to longitudinally describe peripheral oxygen saturation, cerebral oxygen saturation, splanchnic oxygen saturation and regional lung ventilation in extremely low birth weight infants with or without reintubation during the 7 days post extubation.

The application of this multimodal monitoring approach using both clinical and physiological data during the postextubation period will help by making the assessment of clinical stability more comprehensive, more objective, more accurate, more standardized, and more reflective of important end-organ function. Thus, the proposed multimodal monitoring could lead to more informed decisions about reintubation and more individualized treatment plans during this critical period, hence potentially leading to better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1000g and gestational age < 28+0 weeks,
* Received mechanical ventilation within the first 72h of life,
* Undergoing their first planned extubation within the first 6 weeks of life.

Exclusion Criteria:

- Congenital anomalies and congenital heart disorders.

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 20 extremely low birth weight preterm infants admitted to the neonatal intensive care unit at the Montreal Children's Hospital and Centre Hospitalier Universitaire Sainte-Justine.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 168 hours
  To evaluate the time frame needed to recruit patients and percentage of eligible infants recruited
Consent rate | 168 hours
  To evaluate the percentage of eligible infants consented
Acceptability of the multimodal monitoring approach | 168 hours
  Acceptability of the multimodal monitoring approach will be evaluated using short anonymous surveys distributed to parents, bedside nurses, and attending clinicians participating in the study.

SECONDARY OUTCOMES:
To describe longitudinal peripheral blood oxygen saturation patterns for infants with and without reintubation during the 7 days post-extubation | 168 hours
  The variable will be longitudinally described and graphically displayed using mean (standard deviation), median (interquartile range), or number (percentage) for the hour pre-extubation and for each 24-hour bin post-extubation, and compared between infants requiring reintubation and those not requiring reintubation during the 7 days after extubation.
To describe longitudinal cerebral oxygen saturation patterns for infants with and without reintubation during the 7 days post-extubation | 168 hours
  The variable will be longitudinally described and graphically displayed using mean (standard deviation), median (interquartile range), or number (percentage) for the hour pre-extubation and for each 24-hour bin post-extubation, and compared between infants requiring reintubation and those not requiring reintubation during the 7 days after extubation.
To describe longitudinal splanchnic oxygen saturation patterns for infants with and without reintubation during the 7 days post-extubation | 168 hours
  The variable will be longitudinally described and graphically displayed using mean (standard deviation), median (interquartile range), or number (percentage) for the hour pre-extubation and for each 24-hour bin post-extubation. Repeated measures one-way ANOVA or Friedman test will be used to evaluate for differences in the variables over time.
To describe regional lung ventilation from the immediate pre-extubation period until 72-96 hours post-extubation. | 96 hours
  The variable will be longitudinally described and graphically displayed using mean (standard deviation), median (interquartile range), or number (percentage) for the hour pre-extubation and for each 24-hour bin post-extubation. Repeated measures one-way ANOVA or Friedman test will be used to evaluate for differences in the variables over time.

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Shalish, MD, PhD, Principal Investigator — McGill University Health Center/Montreal Children's hospital
Locations (2):
- Canada (2):
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No